CLINICAL TRIAL: NCT05650944
Title: Department of Infectious Disease and Clinical Microbiology
Brief Title: How Important Are Hematological Parameters in the Prognosis of Severe Covid-19 Patients?
Status: Completed | Type: Observational
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Ramazan Gozukucuk, Principal Investigator, Hisar Intercontinental Hospital
Other Study IDs: HisarIH-125
Record Dates: First submitted 2022-12-02; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: Hemogram; NLR; MPV/PLT; MPV/PCT
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 Survivor groups: Covid-19 survivor groups are hematological parameters
  Interventions: Diagnostic Test: Hemogram
- Covid-19 Non-survivor groups: Hematological parameters in patients with severe COVID-19 who have died.
  Interventions: Diagnostic Test: Hemogram

INTERVENTIONS:
Diagnostic Test: Hemogram — Sysmex XN-1000 hematological analyzer

SUMMARY:
It is aimed to reveal the treatment and prognostic values by evaluating the differences in hematological parameters and indices, especially in dead Covid-19 cases.

Material Method: It is planned to retrospectively examine the hemogram parameters of 125 male, 44 female and 169 critical Covid-19 patients hospitalized between 01.03.2020 and 31.12.2021. Subjects were divided into 2 groups as deceased (77) and living (92) patients according to demographic data such as age and gender.

Statistical evaluation: All analyzes were SPSS 25.0, Kolmogorov Smirnov test was used to determine distribution, median and interquartile range (Tukey's Hinges Percentile) were used to summarize variables. The differences between the Independent-Samples Mann Whitney U Test and the data of the patient groups and the optimal cut-off values, sensitivity and specificity values will be determined by ROC analysis. It will be considered statistically significant when the p value is below 0.05 (with the two-tailed test)

DETAILED DESCRIPTION:
The aim of this study is to examine the effectiveness of routine laboratory complete blood count parameters and rates as diagnostic and prognostic criteria in severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18
2. Critical patients taken to intensive care
3. The length of stay in the ICU is more than 24 hours

Exclusion Criteria:

1) Patients under 18 years of age (2) Patients with hematological malignancies (3) The length of stay in the ICU is less than 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study had 169 patients in all, including 44 women and 125 males
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Hematological parameters in the prognosis of severe Covid-19 patients. | 2020-2021
  Hemogram values of the deceased and surviving patients participating in the study were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Gozukucuk, Study Chair — Istanbul Galata Universty
Locations (1):
- Hisar Hospital Intercontinental, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After accepted by Journal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Between 1 March 2020 and 31 December 2021
Access Criteria: All of result open accses.